CLINICAL TRIAL: NCT00153010
Title: A Phase II Double-Blind, Randomized, Dose-Ranging, Placebo-Controlled, Multicenter, Safety and Efficacy Evaluation of Three Doses of NS 2330 in Patients With Mild to Moderate Dementia of the Alzheimer's Type
Brief Title: An Evaluation of Three Doses of NS 2330 in Patients With Mild to Moderate Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1198.52; NCT00055406 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Tesofensine

INTERVENTIONS:
Drug: NS 2330 (Tesofensine)

SUMMARY:
Objectives: The objective of this study will be to determine the safety, tolerability, drug blood levels, and efficacy of each of three doses of NS 2330 (Tesofensine) given once daily compared with placebo in patients with mild to moderate Dementia of the Alzheimer's Type.

ELIGIBILITY:
INCLUSION CRITERIA

Patients may be included in this study if they meet all of the following criteria:

1. Male, and female without child bearing potential between 40 and 85 years of age, inclusive. Women who have been postmenopausal for less than 2 years must have a negative pregnancy test at screening.
2. Diagnosis of probable mild to moderate Dementia of the Alzheimer's Type as defined by National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS ADRDA) guidelines.9
3. Mini-Mental State Examination (MMSE) score of 10-24 and Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) score greater than 12 at screening.
4. Modified Hachinski Scale10 score no greater than 4.
5. Central nervous system imaging (CT or MRI scan of brain) compatible with Dementia of the Alzheimer's Type within the past year (also see exclusion criteria).
6. Exhibits reliability and physiologic capability sufficient to comply with all protocol procedures. Patient must be familiar with and fluent in English (i.e., sufficient to complete all study assessments from the language perspective).
7. Patients and/or a legal representative and their caregivers must have given informed consent. The legal representative and caregiver may be the same person.
8. Patient must have a reliable caregiver that is in frequent or daily contact with the patient, who will accompany the patient to the office and who will monitor the administration of prescribed medications. The caregiver will be able to communicate in English and be willing to comply with protocol requirements.

EXCLUSION CRITERIA

Patients must be excluded from this study if they meet any of the following criteria:

1. Secondary disorders inducing dementia such as neurosyphilis, craniocerebral trauma (CT/MRI), hyperthyroidism, or folic acid deficiency.
2. History of malignancy within 3 years, except for basal cell carcinoma.
3. History or diagnosis of symptomatic and/or unstable/uncontrolled:

   * Cardiovascular illnesses such as chronic congestive heart failure (with or without edema), arrhythmias, labile hypertension, ischemic heart disease, myocardial infarction (with residual angina), orthopnea, conduction defects (ECG), or other heart disease classified NYHA III or IV.
   * Liver disease such as cirrhosis, hepatitis B, hepatitis C, or primary or metastatic neoplasm.
   * Gastrointestinal disorder such as GI bleeding, malabsorption syndromes, post-gastrectomy, or active peptic ulcer disease.
   * Renal disease (primary or secondary) such as chronic renal failure (CLCR < 30 mL/min).
   * Endocrine disease such as diabetes mellitus or hypothyroidism.
   * Neurological disease (other than Dementia of the Alzheimer's Type such as Huntington's disease, Parkinson's disease, encephalitis, epilepsy, stroke, or multiple sclerosis) and psychiatric disorders such as schizophrenia, major depression, or mental retardation.
   * Significant pulmonary disease predisposing to hypoxia.
   * Immunological disorder such as clinically significant allergies, Lupus erythematosis, or scleroderma.
   * Hematological disease (regardless of cause) such as refractory anemia or refractory myelosuppression.
   * Organ system diseases which, in the opinion of the investigator, would impact on the primary and secondary endpoints of the trial such as dehydration (hematocrit >48%) or hypothyroidism.
4. Significant history of drug dependence or abuse (including alcohol, as defined in DSM IV or in the opinion of the investigator) within two years, or a positive urine drug screen for cocaine, heroin, or marijuana.
5. HIV positive.
6. Presence of Hepatitis C antibody.
7. Planned elective surgery requiring general anesthesia or hospitalization for more than 1 day during the study period.
8. Previous participation in any NS 2330 study.
9. Use of any investigational drug or procedure within 30 days before randomization.
10. Use of any drug within 14 days prior to randomization unless:

    * the dose of the drug and the condition being treated have been stable for at least 30 days and are expected to remain stable during the study
    * neither the drug nor the condition being treated is expected to interfere with the study endpoints.
11. Treatment with donepezil, galantamine, rivastigmine, or tacrine, is prohibited within 6 weeks before randomization.
12. Treatment with drugs that inhibit CYP 450 3A4 (see Appendix II for a list of relevant drugs.) If they are needed under emergency conditions, the patient should discontinue the trial.
13. Treatment with antipsychotics/neuroleptics is prohibited for 8 weeks prior to randomisation (see listing Appendix II).
14. Treatment with monoamine oxidase inhibitors is prohibited for 8 weeks prior to randomization.
15. Treatment with selective serotonin reuptake inhibitors is prohibited for 6 weeks prior to randomization.
16. Tricyclic antidepressants and antihistamines are prohibited for 4 weeks prior to randomization.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2003-02; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Changes in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | week 0, 4, 9, 14 and 20

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change | weeks 0 and 14
Alzheimer's Disease Cooperative Study-Activities of Daily Living | weeks 0, 4, and 14
Neuropsychiatric Inventory | weeks 0, 4, and 14
Mini-Mental State Examination | weeks 0 and 14
ADAS-Cog Extension | weeks 0, 4, 9, 14 and 20
ADAS-Cog total score including Extension | weeks 0, 4, and 14
types and frequencies of adverse events | 20 weeks
proportion of patients discontinued from the trial because of adverse events | 20 weeks
changes from baseline in vital signs | 20 weeks
changes from baseline in laboratory measurements | 20 weeks
changes from baseline in ECG readings | 20 weeks
comparison of study groups for drug plasma concentrations | weeks 0, 4, 9, 14 and 20
population PK parameters | Weeks 0, 4, 9, 14 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (87):
- United States (80):
  - Pivotal Research Center, Mesa, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Xenoscience, Phoenix, Arizona
  - Boehringer Ingelheim Investigational Site, Berkeley, California
  - California Clinical Trials Medical Group, Culver City, California
  - Margolin Brain Institute, Fresno, California
  - Care@ Granada Hills Community Hospital, Granada Hills, California
  - Optimum Health Services, La Mesa, California
  - Optimum Health Services, Oceanside, California
  - Southwest Institute for Clinical Research, Rancho Mirage, California
  - Health Quest Clinical Trials, San Diego, California
  - Institute on Aging Research Center, San Francisco, California
  - Torrance Clinical Research, Torrance, California
  - Associated Neurologists PC - Danbury, Danbury, Connecticut
  - Center for Geriatric & Adult Psychiatry, Hamden, Connecticut
  - Neurology Associates PA, Wilmington, Delaware
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Florida
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Neurologic Consulting/PA, Fort Lauderdale, Florida
  - Clinical Physiology Associates Study Center, Fort Meyers, Florida
  - Berma Research Group, Hialeah, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Baumel-Eisner Neuromedical Institute, Miami, Florida
  - Miami Jewish Home and Hospital for the Aged, Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Magnolia Research Group, Ocala, Florida
  - Memory Disorder Clinic, Pompano Beach, Florida
  - Boehringer Ingelheim Investigational Site, Tampa, Florida
  - USF Suncoast Gerontology Center, Tampa, Florida
  - Palm Beach Neurology/Premier Research Institute, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Peryam and Kroll Healthcare Research, Chicago, Illinois
  - LaGrange Hospital, LaGrange, Illinois
  - Agewell, Ltd., Indianapolis, Indiana
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Hartford Research Group, Florence, Kentucky
  - Associates in Neurology-Research, Lexington, Kentucky
  - Louisiana State University Medical Center, New Orleans, Louisiana
  - Attn: M. Lannom, RN, MS, Sharon, Massachusetts
  - Future Care Studies, Springfield, Massachusetts
  - Saginaw Cooperative Hosp. Inc./ Internal medicine, Saginaw, Michigan
  - North Michigan Neurology, Traverse City, Michigan
  - University of Missouri, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Atlantic Coast Research, Toms River, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Neurological Associates of Albany, Albany, New York
  - Upstate Clinical Research, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - Eastside Comprehensive Medical Services, New York, New York
  - Social Psychiatry Research Institute, New York, New York
  - The Jewish Home and Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Triangle Medical Research, Lexington Road, North Carolina
  - Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - North Coast Clinical Trials, Inc., Beachwood, Ohio
  - Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neurology Center of Ohio, Toledo, Ohio
  - Linden Research Consultants, Oklahoma City, Oklahoma
  - Pahl Brain Associates, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigators, Inc., Eugene, Oregon
  - PRO Research, Eugene, Oregon
  - Attn: Valerie MacDonald, Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Crosswords Counseling and Consulting Associates, Moon Township, Pennsylvania
  - Pearl Clinical Research, Inc., Norristown, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital Dept. of Neurology, Providence, Rhode Island
  - Medical Univ. of South Carolina, Alzheimer's Research, North Charleston, South Carolina
  - Psychiatric Consultants, Nashville, Tennessee
  - Baylor College of Medicine VA Medical Center, Houston, Texas
  - University of Texas Medical Science Institute, Houston, Texas
  - Caprock Clinical Trials Center, Lubbock, Texas
  - Integra Clinical Research, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - The Memory Clinic/Southwestern Vermont Medical Center, Bennington, Vermont
  - UVA Dept. of Neurology, Charlottesville, Virginia
  - Independent Psychiatric Consultants, Waukesha, Wisconsin
- Canada (7):
  - Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - Infectious Disease, Moncton, New Brunswick
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Clinical Research Consultant Group, Beaconsfield, Quebec
  - Boehringer Ingelheim Investigational Site, Greenfield Park, Quebec
  - Pasqua Hospital, Regina, Saskatchewan